CLINICAL TRIAL: NCT03709992
Title: Trospium Chloride vs Tamsulosin in Treatment of Ureteral Stent Related Symptoms: A Randomized Controlled Trial
Brief Title: Trospium Chloride vs Tamsulosin in Treatment of Ureteral Stent Related Symptoms:
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of COVID-19 Crisis
Sponsor: Mansoura University (Other)
Collaborators: Amiri Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmed R. EL-Nahas, Professor of Urology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Trospium vs Tamsulosin
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Ureter Stone; Quality of Life; Ureter Obstruction
Keywords: ureteral stent; USSQ; Tamsulosin; Trospium Chloride
MeSH Terms: conditions — Ureterolithiasis; Ureteral Obstruction | interventions — trospium chloride; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trospium (Active Comparator): Patients will receive 30 mg of Trospium chloride tablet twice daily
  Interventions: Drug: Trospium Chloride
- Tamsulosin (Active Comparator): Patients will receive 0.4 mg of Tamsulosin tablet once daily
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Trospium Chloride — 30 mg of Trospium chloride tablet twice daily
  Other Names: Spasmix
  Arms: Trospium
Drug: Tamsulosin — 0.4 mg of Tamsulosin tablet once daily
  Other Names: Omnic
  Arms: Tamsulosin

SUMMARY:
This study will be conducted to compare the efficacy and safety of Trospium chloride versus Tamsulosin for treatment of ureteral stent related symptoms.

DETAILED DESCRIPTION:
Eligible patients will be randomized to one of the two treatment groups. Group 1 patients will receive 30 mg of Trospium chloride tablet twice daily, while group 2 patients will receive 0.4 mg of Tamsulosin tablet once daily, until the stent is removed. Ureteral Stent Symptoms Questionnaire (USSQ) will be used to evaluate the symptoms of the patients with DJ stent after 2 weeks of inserting the stent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with double "J" (DJ) stent after ureteroscopy or for drainage of obstructed kidney

Exclusion Criteria:

1. Patients with hypersensitivity to either Trospium chloride or Tamsulosin
2. Patients with complications after DJ insertion (such as fever, hematuria, perforation, stent migration).
3. Patients receiving alpha blockers or anticholinergic medications for any other reason.
4. Patients with history of orthostatic hypotension.
5. Pregnant or breastfeeding females.
6. Patients with hepatic impairment (Child-Pugh score >9).
7. Patients with severe renal impairment with creatinine clearance of less than 15 mL/min.
8. Patients with narrow-angle glaucoma.
9. Patients with history of urinary retention or gastric retention.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Ureteral Stent Symptoms Questionnaire (USSQ) score | 14 days
  Quantitative assessment of quality of life score

SECONDARY OUTCOMES:
Adverse events | 14 days
  Assessment of side effects of the drug used

CONTACTS AND LOCATIONS:
Overall Officials: Abdullatif AL-Terki, MD, Study Chair — Amiri Hospital - Kuwait
Locations (1):
- Ahmed R EL-Nahas, Al Mansurah, Kuwait, Egypt

IPD SHARING:
Plan to Share IPD: No